CLINICAL TRIAL: NCT02870400
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of Intravenously and Subcutaneously Administered REGN2477 in Healthy Women Not of Childbearing Potential
Brief Title: A Study to Examine the Safety and Tolerability of Single Ascending Doses of REGN2477
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R2477-HV-1525
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- REGN2477 (Experimental): Cohorts 1 - 5 will receive REGN2477
  Interventions: Drug: REGN2477
- Placebo (Experimental): Cohorts 1 - 5 will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN2477 — Participants will receive ascending doses of REGN2477
  Arms: REGN2477
Drug: Placebo — Participants will receive matching placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of single ascending doses of REGN2477 in healthy women not of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women not of childbearing potential between 18 and 65 years of age, with no significant health issues or clinically significant abnormal laboratory findings
2. A body mass index (BMI) between 18 to 30 kg/m2, inclusive
3. Provide a signed informed consent

Exclusion Criteria:

1. Significant illness or history of significant illness
2. Clinically significant abnormal CBC, clinical chemistry, and urine analysis at screening
3. Current smoker or former smoker who has stopped smoking within 3 months prior to screening
4. Positive urine drug test results during screening, or history of drug or alcohol abuse
5. Donation or loss of, blood within 8 weeks prior to screening, or plasma up to 14 days prior to screening
6. History of diabetes
7. Abnormal blood pressure (BP)
8. History of gynecological disorders or malignancies; history of breast malignancies; or history of benign gynecological or breast lesions that require medical treatment or follow up
9. Reduced renal function
10. Known history of chronic hepatitis or HIV
11. Clinically significant ECG abnormalities
12. Participation in any clinical research study within 30 days, or 5 halflives, of the study drug, whichever is greater, or for longer periods per regional requirements, prior to the screening visit
13. Exposure to any biological drugs within 3 months of the screening visit (the name of the drug and duration of previous exposure will be recorded). Vaccination within 4 weeks of screening visit.
14. History of hypersensitivity reactions to vaccines or other biologics
15. History of hypersensitivity to doxycycline or other tetracycline antibiotics
16. History of osteoporosis requiring osteoporosis treatments such as PTH, bisphosphonates, and denosumab
17. Subject using hormone replacement therapy or thyroid replacement therapy will be excluded, unless they have been on stable doses of such therapy for at least 6 months and will remain on the same stable dose through the duration of the trial
18. Use of systemic glucocorticoids, including oral glucocorticoids, for more than 10 days, within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) through day 113 in participants treated with REGN2477 | Day 1 to Day 113

SECONDARY OUTCOMES:
Pharmacokinetic profile of REGN2477, assessed via serum concentrations of REGN2477 over time | Day 1 to Day 113
Immunogenicity of REGN2477, as determined by the presence or absence of Anti-drug antibody (ADA) to REGN2477 over time | Day 1 to Day 113

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Antwerp, Belgium